CLINICAL TRIAL: NCT07306598
Title: [18F]NIDF PET Imaging in Tau-related Diseases
Status: Recruiting | Type: Observational
Sponsor: Tianjin Medical University (Other)
Collaborators: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Shaobo Yao, PhD, Prof., Tianjin Medical University
Other Study IDs: TJMUGH-13
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Neurodegenerative Disease; Alzheimer s Disease; Tauopathies
Keywords: PET/CT; Alzheimer's disease; Tau pathologies; Tauopathies
MeSH Terms: conditions — Neurodegenerative Diseases; Tauopathies; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy participants: Participants will receive a single intravenous bolus injection of 10 ± 3 mCi of [18F]NIDF followed by a PET/CT scan.
- Patients with cognitive impairment: Participants will receive a single intravenous bolus injection of 10 ± 3 mCi of [18F]NIDF followed by a PET/CT scan.

SUMMARY:
In the field of diagnosing brain neurodegenerative diseases, it is now a well-established practice to inject positron-emitting tracers into the human body. These tracers bind to specific target proteins, allowing their distribution to be visualized via PET imaging. Currently, several research groups worldwide are engaged in developing and clinically validating their own tau imaging agents.

This clinical research project aims to visualize abnormal tau pathology in the living human brain using [18F]NIDF PET imaging. [18F]NIDF is a 2-arene-azaindole-based tracer that offers stronger binding affinity to tau neurofibrillary tangles and reduced non-specific/off-target binding compared to existing tau-PET imaging agents. The study primarily focuses on evaluating the safety and diagnostic efficacy of [18F]NIDF PET imaging in human subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 90 years old;
2. No gender limitation;
3. Clinical diagnositic rerults supported the diagnosis of neurodegeneration, and there was no evidence of other neurological diseases;
4. Healthy participants or patients with probable Alzheimer's disease or with dementia due to other causes;
5. Informed consent signed in person by the subject or his legal guardian or caregiver.

Exclusion Criteria:

1. Has allergy to [18F]NIDF or any of its excipients;
2. Incapable of providing written informed consent or lacking a legally authorized representative (LAR) to provide informed consent ;
3. Unwilling or unable to undergo PET scans tracer injections;
4. Any condition that, in the Investigator's opinion, could increase the risk to the participant, limit the participant's ability to tolerate the research procedures, or interfere with the collection/analysis of the data (e.g., renal or liver failure, advanced cancer);
5. Received an experimental drug or device within 1 month (whose efficacy or safety is unclear);
6. Have other serious neurological disorders, or gastrointestinal, cardiovascular, liver, kidney, blood system, tumor, endocrine, respiratory, immune deficiency, and other serious diseases;
7. Women who are currently pregnant or breastfeeding.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Researchers look for people who fit a certain description, called eligibility criteria. Some examples of these criteria are a person's general health condition or prior treatments.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety Assessment | From time of injection up to 7 days post-injection
  The incidence of adverse events assessed by the investigator as related to the [18F]NIDF injection. Systematically collect and assess all adverse events within 7 days post-injection through physical examinations, vital signs monitoring, clinical laboratory tests (complete blood count, hepatic and renal function). All events will be graded for severity according to the Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
The Biodistribution of [18F]NIDF in subjects | At the time of the single [18F]FT8 PET/CT scan (Day 1)
  Semi-quantitatively evaluate the tracer's uptake in the interest brain regions, like cortical cortex, hippocampus and cerebellum, by measuring the Standard Uptake Value (SUV) or % inject dose per volum (%ID/cc).

SECONDARY OUTCOMES:
Diagnostic Performance | From enrollment to the end of PET/CT sacns at 2 weeks
  Diagnostic performance including sensitivity, specificity, accuracy. Quantification of [18F]NIDF uptake in different brain regions (e.g., amygdala, temporal lobe, hippcampus) using the Standardized Uptake Value (SUV). This measurement will be performed on the PET/CT scans acquired at a specified time. The outcome will be reported as the SUV in both two groups.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No